CLINICAL TRIAL: NCT05186454
Title: Multimodal Intrathecal Analgesia for Cesarean Section
Brief Title: Postoperative Pain Control by Use of Many Drugs in Small Doses Intrathecally
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fouad Soliman, Lecturer of Anesthesia and ICU, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2008
Record Dates: First submitted 2021-12-26; First posted 2022-01-11 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Post Operative Pain
Keywords: Intrathecal morphine, midazolam, dexamethasone, cesarean section
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; Bupivacaine; Dexamethasone; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphine (Active Comparator): Patients will receive 10-12.5 mg bupivacaine and 1 ml containing 200 µg of morphine intrathecally.
  Interventions: Drug: Morphine Sulfate; Drug: Bupivacaine
- Multimodal (Active Comparator): Patients will receive 10-12.5 mg bupivacaine and 1 ml containing 2 mg dexamethasone, 50 µg morphine, and 500 µg midazolam intrathecally
  Interventions: Drug: Bupivacaine; Drug: dexamethasone, morphine, midazolam

INTERVENTIONS:
Drug: Morphine Sulfate — analgesia
  Other Names: bupivacaine
  Arms: Morphine
Drug: Bupivacaine — Analgesia
Drug: dexamethasone, morphine, midazolam — 1 ml containing 2 mg dexamethasone, 50 µg morphine, and 500 µg midazolam
  Arms: Multimodal

SUMMARY:
Cesarean section is one of the painful operations that require adequate postoperative analgesia. Patients are divided into two groups: Multimodal (DMM) group ( 30 patients): patients will receive spinal anesthesia with 10-12.5 mg bupivacaine and 1 ml containing 2 mg dexamethasone, 50 µg morphine, and 500 µg midazolam.

Morphine (M) group (30 patients): patients will receive spinal anesthesia with 10-12.5 mg bupivacaine and 1 ml containing 200 µg morphine

ELIGIBILITY:
Inclusion criteria:

* ASA I-II
* Age 20-40 years.
* Pregnant women with living fetus.
* Body mass index 20- 35 kg/m2.

Exclusion criteria:

* Patient refusal.
* Age < 20 or > 40 years
* Body mass index < 20 or > 35.
* Contraindication to spinal anesthesia (severe mitral or aortic stenosis, coagulopathy, Systemic or local infection, increased intracranial pressure and hypovolemia).
* Placental abnormalities: placental abruption, placenta previa or accrete.
* Allergy to drugs used in the study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-23 (Actual); Primary Completion 2022-02-10 (Estimated); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
1st analgesic requirement | 24 hours
  The first time of supplemental analgesic need postoperatively

SECONDARY OUTCOMES:
Analgesic consumption | 24 hours
  Total analgesic consumption
Post operative pain | 24 hours
  Visual Analog Scale(0-10 with 0 is no pain and 10 is maximum intolerable pain)
Side effects | 24 hours
  1. Pruritus (assessed the number of patients suffering from pruritus and grading the degree as follow:Mild= Itching is a minor concern, Moderate = Itching is a primary concern, but bearable,Severe= Unbearable; patient need anti-histaminic treatment.
  2. Nausea and/or vomiting(assessed on 4 grade scales:
  0= no symptoms present, 1 =mild nausea with no need for pharmacological treatment, 2= moderate nausea that required treatment (ondansetron 4 mg), 3= severe nausea that is resistant to treatment).
  3-Sedation (assessed on 4 grade scale: 1-awake and alert, 2 -slightly drowsy, easily aroused, 3 -drowsy, drifts off to sleep during conversation, 4 -somnolent, minimal, or no response to physical stimulation).
  4- Respiratory depression whether present or not(Respiratory depression was defined as a respiratory rate ≤10/min.)

CONTACTS AND LOCATIONS:
Locations (1):
- Fouad Soliman, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No